CLINICAL TRIAL: NCT06972888
Title: A Multicenter, Randomized, Double-blind, Parallel-group, Placebo-controlled Phase II Clinical Study to Evaluate the Efficacy, Safety, and Pharmacokinetic Profile of AC-201 Tablets in Subjects With Moderate-to-severe Plaque Psoriasis
Brief Title: A Phase II Clinical Study of AC-201 Tablets in Subjects With Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Accro Bioscience (Suzhou) Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AC201-003
Record Dates: First submitted 2025-05-07; First posted 2025-05-15 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — diacerein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1: AC-201 Dose 1 (Experimental): Subjects will receive AC-201 Dose 1 as tablets orally twice daily from Week 0 through W12
  Interventions: Drug: AC-201
- Group 2: AC-201 Dose 2 (Experimental): Subjects will receive AC-201 Dose 2 as tablets orally twice daily from Week 0 through W12
  Interventions: Drug: AC-201
- Group 3: AC-201 Dose 3 (Experimental): Subjects will receive AC-201 Dose 3 as tablets orally twice daily from Week 0 through W12
  Interventions: Drug: AC-201
- Group 4: Placebo (Experimental): Subjects will receive matching placebo as tablets orally twice daily from Week 0 through W12
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AC-201 — AC-201 tablets will be administered orally
  Arms: Group 1: AC-201 Dose 1; Group 2: AC-201 Dose 2; Group 3: AC-201 Dose 3
Drug: Placebo — Matching placebo tablets will be administered orally.
  Arms: Group 4: Placebo

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of AC-201 tablets compared with placebo in subjects with moderate-to-severe plaque psoriasis

DETAILED DESCRIPTION:
AC-201 is a highly selective dual inhibitor of TYK2 and JAK1, which are targeting the signal transduction of a variety of cytokines in psoriasis. This study is to evaluate the efficacy and safety of AC-201 tablets in subjects with moderate-to-severe plaque psoriasis. The efficacy will be determined by the superior percentage of subjects achieved Psoriasis Area and Severity Index (PASI) 75 (greater than or equal to 75% improvement in PASI) compared with placebo. The treatment of AC-201 will be up to 12 weeks and followed by a 4-week safety follow-up, and total duration will be up to 16 weeks. Adverse Events, clinical laboratory assessments, electrocardiograms (ECGs), vital signs, physical examinations, concomitant medications will be monitored throughout the study. Meanwhile, pharmacokinetics and pharmacodynamics will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

-Stable plaque psoriasis (defined as no morphological or severity changes for ≥ 6 month) and meet the following disease severity at screening and baseline: Total PASI score ≥ 12, and Total sPGA ≥ 3, and Total BSA ≥ 10%

-Candidate for phototherapy or systemic treatment for plaque psoriasis

Exclusion Criteria:

* Other form of psoriasis (e.g., erythrodermic, pustular or guttate)
* Current or history for drug-induced psoriasis (e.g., psoriasis induced by beta blockers, calcium channel blockers, antimalarial drugs, or lithium)
* History or risk of tuberculosis (TB)
* Have received TYK2 inhibitor and lack of efficacy deemed by investigator
* Topical medications/treatments for psoriasis within 2 weeks prior to administration of any study medication
* Systemic medications/treatments for psoriasis within 4 weeks prior to administration of any study medication
* Has received biological treatment (e.g., anti-TNFα, anti-IL12/23, anti-IL17) for psoriasis less than 5 half-lives of treatment prior to administration of any study medication

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2024-04-23 (Actual); Primary Completion 2025-03-07 (Actual); Study Completion 2025-04-28 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects achieved Psoriasis Area Severity Index (PASI) 75 at Week 12 | Week 12
  Percentage of subjects achieved PASI 75 (greater than or equal to 75% improvement from baseline in PASI) at Week 12 will be reported. The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: head, trunk, upper, and lower extremities. Each of these areas is assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90% to 100% involvement), and for erythema, induration, and scaling, which are each rated on a scale of 0 (none) to 4 (severe). The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease.

SECONDARY OUTCOMES:
Change from baseline in Psoriasis Area Severity Index (PASI) score at Week12 | Baseline and Week 12
  Change from baseline in PASI score at Week 12 will be reported. The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: head, trunk, upper, and lower extremities. Each of these areas is assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90% to 100% involvement), and for erythema, induration, and scaling, which are each rated on a scale of 0 (none) to 4 (severe). The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease.
Percentage of subjects achieved Psoriasis Area Severity Index (PASI) 90 at Week 12 | Week 12
  Percentage of subjects achieved Psoriasis Area Severity Index (PASI) 90, (greater than or equal to 90% improvement from baseline in PASI) at Week 12 will be reported. The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: head, trunk, upper, and lower extremities. Each of these areas is assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90% to 100% involvement), and for erythema, induration, and scaling, which are each rated on a scale of 0 (none) to 4 (severe). The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease.
Percentage of subjects achieved static Physician Global Assessment (sPGA) of 0 or 1 (sPGA 0/1) at Week 12 | Week 12
  Percentage of subjects achieved sPGA 0/1 at Week 12 will be reported. The sPGA is a 5-point scale of an average assessment of all psoriatic lesions based on erythema, scaling, and induration. The average of the 3 scales, rounded to the nearest whole number, is the final sPGA score. The sPGA score ranges from 0 to 5 (0 = clear, with no evidence of plaque elevation, erythema, or scale, and 5 = severe induration, erythema, and scaling).
Change from baseline in Body Surface Area (BSA) at Week 12 | Baseline and Week 12
  Change from baseline in BSA at Week 12 will be reported. BSA is a commonly used measure of extent of skin disease. It is defined as the percentage of surface area of the body involved with the condition being assessed.
Number of subjects with Adverse Events | Up to Week 16
  An Adverse Event (AE) is defined as any new untoward medical condition or worsening of a pre-existing medical condition following or during exposure to an investigation product, whether or not considered causally related to the product.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of China Medical University, Shenyang, China

IPD SHARING:
Plan to Share IPD: No